CLINICAL TRIAL: NCT06061640
Title: The Potential Value and Impact of Diagnostic Biomarkers for MAFLD Using Machine Learning Methods
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-KL-202-01
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Metabolic Dysfunction-associated Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: MAFLD patients
- control group: health people

SUMMARY:
This is a case-control study that aims to build a predictive model for MAFLD based on machine learning.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated fatty liver disease (MAFLD) also known as non-alcoholic fatty liver disease (NAFLD), is one of the most prevalent liver diseases worldwide with high prevalence and economic burden, which affects 25% of global adult population. Despite extensive research on understanding the inner pathophysiology of MAFLD, it still keep growing with no approval therapy. Therefore, preventive measures are particularly important in diagnosing MAFLD. So far the liver biopsy is still the gold standard for diagnosis of MAFLD, however considering the invasive process and potential risks, it still has low acceptance for asymptomatic patients, thus non-invasive methods are necessary for this reason.

The purpose of this study is to establish a prediction model to identify MAFLD patients, which can accurately predict whether the participants have MAFLD according to the relevant metabolic indicators of the participants, without the need for invasive examinations such as tissue biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 75 years;
2. meeting the diagnostic criteria of MAFLD;
3. no other organic lesions were found in imaging examination;
4. willing and able to sign informed consent.

Exclusion Criteria:

1. significant drinking history (weekly alcohol consumption ≥ 140g for male, or weekly alcohol consumption ≥ 70g for female);
2. presence of evidence for having hepatic steatosis, viral hepatitis, history of hepatic cancer, drug-induced liver injury, liver cirrhosis and other liver and biliary tract diseases;
3. major organ malfunction, severe systemic illnesses, mental health issues, or inability to complete examination;
4. pregnant or pregnancy planning female;
5. missing of important clinical data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese participants age 18 years or older diagnosed with MAFLD on imaging and healthy volunteers without MAFLD.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under cure | 2022-2024
  Area under cure(AUC) was defined as the area enclosed by the coordinate axis under the receiver operating characteristic curve, with values ranging from 0.5 to 1.0. The closer the AUC is to 1.0, the higher the authenticity of the detection method; the closer to 0.5, the lower the authenticity of the detection method; when equal to 0.5, the authenticity is the lowest and has no application value.

SECONDARY OUTCOMES:
Accuracy | 2022-2024
  The proportion of the number of correctly classified samples to the total number of samples.
Precision | 2022-2024
  The proportion of data that is actually positive among the data that is determined to be positive.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Clinical Medical College of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China